CLINICAL TRIAL: NCT01949688
Title: Phase I/II Study Using Epitope Peptide Restricted to HLA-A*24 or HLA-A*02 in Patients With Advanced Solid Tumors That Are Refractory to Standard Therapy
Brief Title: Safety and Efficacy Study of Epitope Peptide To Treat HLA-A*24 or A*02-positive Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shiga University (Other)
Collaborators: Tokyo University (Other)
Responsible Party: Principal Investigator, Yataro Daigo, Professor, Shiga University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUMS-22-15; 22-15 (Other: Shiga University)
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Solid Tumors
MeSH Terms: interventions — HLA-A*24:02 antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HLA-A*2402 restricted peptides (Experimental): HLA-A*2402 restricted peptides with adjuvant
  Interventions: Biological: HLA-A*2402 or A*0201 restricted peptides
- HLA-A*0201 restricted peptides (Experimental): HLA-A*0201 restricted peptides with adjuvant
  Interventions: Biological: HLA-A*2402 or A*0201 restricted peptides

INTERVENTIONS:
Biological: HLA-A*2402 or A*0201 restricted peptides — Open Label, Non-Randomized, Safety/Efficacy study:
  1. HLA-A*2402-positive patients will be vaccinated subcutaneously once a week with HLA-A*2402 restricted peptides for VEGF-R1 and VEGF-R2 with adjuvant.
  2. HLA-A*0201-positive patients will be vaccinated subcutaneously once a week with HLA-A*0201 restricted peptides for VEGF-R1 and VEGF-R2 with adjuvant.

SUMMARY:
In this study, the investigators examine using a combination of two types of HLA-A*2402 (or HLA-A*0201)-restricted epitope peptides, which were derived from VEGF-R1 and VEGF-R2 the safety, immunogenicity, and antitumor effect of vaccine treatment for advanced solid tumor patients who are refractory to standard therapy.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability, immune response and clinical efficacies of HLA-A*2402 or HLA-A*0201 restricted epitope peptides (VEGF-R1 and VEGF-R2) emulsified with Montanide ISA 51 for advanced solid tumors.

In this phase I/II trial, the investigators examine using a combination of the two peptides the safety, immunogenicity, and antitumor effect of vaccine treatment for HLA-A*2402 or HLA-A*0201-positive advanced solid tumor patients who are refractory to standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced solid tumors that are refractory to standard therapies or that cannot be treated with those due to medical reason.
2. ECOG performance status 0-1
3. Age between 20 to 85
4. Clinical efficacy can be evaluated by some methods
5. No prior chemotherapy, radiation therapy, hyperthermia or immunotherapy within two weeks
6. Life expectancy > 3 months
7. Laboratory values as follows 1500/mm3 < WBC < 10000/mm3 Platelet count > 75000/mm3 15% < Lymphcyte fraction Asparate transaminase < 3 X cutoff value Alanine transaminase < 3 X cutoff value Total bilirubin < 3 X cutoff value Serum creatinine < 2X cutoff value
8. HLA-A*2402 or HLA-A*0201
9. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Active and uncontrolled cardiac disease (i.e. coronary syndromes, arrhythmia)
2. Myocardial infarction within six months before entry
3. Breastfeeding and Pregnancy (woman of child bearing potential)
4. Active and uncontrolled infectious disease
5. Concurrent treatment with steroids or immunosuppressing agent
6. Other malignancy requiring treatment
7. Non-cured traumatic wound
8. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2010-06; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety: the number of adverse events of vaccination therapy. | 2 months
Evaluation of clinical efficacy: Overall survival. | 2 months

SECONDARY OUTCOMES:
Various immunological responses including peptides specific CTL, antigen cascade, regulatory T cells, cancer antigens and HLA levels. | 2 months
Evaluation of clinical efficacy: Progression free survival. | 2 months
Evaluation of clinical efficacy: Tumor markers. | 2 months
Evaluation of clinical efficacy: Objective response rate. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Yataro Daigo, MD, PhD, Principal Investigator — Shiga University
Locations (1):
- Shiga University of Medical Science Hospital, Ohtsu, Shiga, Japan